CLINICAL TRIAL: NCT03101683
Title: Partial Chest Wall Radiation Therapy After Total/Skin Sparing Mastectomy and Immediate Implant-based Reconstruction for Breast Cancer Patients at Increased Risk of Local Recurrence
Brief Title: Radiotherapy After Mastectomy for Breast Cancer Patients at Increased Risk of Local Recurrence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondazione del Piemonte per l'Oncologia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCWRT-01
Record Dates: First submitted 2017-03-03; First posted 2017-04-05 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PCWRT Group (Experimental): Patients with diagnosis of in situ ductal carcinoma (pTis) or invasive breast carcinoma (pT1 and pT2), submitted to NAC sparing mastectomy with prosthetic-based breast reconstruction who have some additional risk factors will receive a partial chest wall radiotherapy
  Interventions: Radiation: Partial chest wall radiation therapy

INTERVENTIONS:
Radiation: Partial chest wall radiation therapy — A dose of 40 Gy in 16 fractions (2.5 Gy per fraction) is delivered in the area at risk of local recurrence (skin and the pectoralis muscles) delineated by surgical clips and 3D-MRI reconstruction for a precise localization of the tumor excised

SUMMARY:
STUDY DESCRIPTION: This is a single-arm study to assess the feasibility, toxicity and cosmetic outcome of partial radiotherapy of the chest wall in breast cancer patients at increased risk of local relapse submitted to nipple-areola complex (NAC) sparing mastectomy and immediate implant-based reconstruction Inclusion criteria

Histologically confirmed diagnosis of in situ ductal carcinoma (pTis) or invasive breast carcinoma (pT1 and pT2), submitted to NAC sparing mastectomy with prosthetic-based breast reconstruction (expander or prosthesis) and:

Group A)

Negative sentinel node dissection or axillary clearance (pN0) and all the following risk factors:

Close (less than 1 mm) or positive (ink on tumor margin) surgical margin in a single breast quadrant Tumor diameter >2 cm Age ≤50 years Group B)

Positive sentinel dissection (pN1a) followed by axillary clearance (or primary axillary clearance) with only 1 positive node and any of the following risk factors:

Close (less than 1 mm) or positive (ink on tumor margin) surgical margin in a single breast quadrant Age ≤50 years Tumor diameter >2 cm Grade 3 histology Lymphovascular invasion HER-2 overexpression/amplification Triple negativity Treatment - Radioterapy The tumor bed is defined by the area at risk (skin and the pectoralis muscles) delineated by surgical clips and 3D-MRI reconstruction for a precise localization of the tumor excised. The clinical target volume (CTV) is defined as the tumor bed with a 1.5 cm margin limited by skin contour.

A dose of 40 Gy is delivered in 16 fractions (2.5 Gy per fraction). For conventional post-mastectomy radiotherapy this moderately hypofractionated schedule is considered feasible and safe (31). Even more so, this schedule should be feasible and safe for a smaller irradiated volume as in the current protocol. Regional nodal irradiation is not considered at our Institution for patients fulfilling the entry criteria of the protocol.

OUTCOME MEASURES Primary To assess feasibility of PCWRT via VMAT-IGRT linac-based or helical Tomotherapy To assess the safety of PCWRT via VMAT-IGRT linac-based or helical Tomotherapy To assess the surgical complication of implant-based breast reconstruction after PCWRT Secondary To assess the cosmetic outcome of implant-based breast reconstruction after PCWRT To assess patients' satisfaction of implant-based breast reconstruction after PCWRT

DETAILED DESCRIPTION:
There is uncertainty on the indications to chest wall irradiation in patients submitted to mastectomy plus immediate implant-based reconstruction with: A) negative axillary nodes and additional risk factors; B) 1-3 positive axillary nodes and no additional risk factors.

The reduction of locoregional recurrences is valuable from a clinical and psychological standpoint and may also translate into a survival advantage. Nevertheless, whole chest wall radiotherapy can be associated with significant toxicity due to irradiation of non-target organs and does significant worsen the cosmetic result of prosthetic-based breast reconstruction (capsular contracture, implant displacement, infection).

Most Institution have adopted NAC sparing mastectomy as standard treatment for non-locally advanced breast cancer patients not amenable to breast conserving surgery. Available literature data, including our own data, suggest that in these patients local recurrence in the NAC area is exceedingly rare, while most local recurrences occur where the original tumor was located.

It is now accepted that, in selected breast cancer patient submitted to breast conserving surgery, accelerated partial breast radiotherapy is associated with similar recurrence rates as compared to whole breast radiotherapy and favorable cosmetic outcomes. Therefore, we hypothesize that partial chest wall radiotherapy of the quadrant where the original tumor was located after NAC sparing mastectomy may be associated with the same reduction of local recurrences while significantly reducing the complications of prosthetic-based breast reconstruction.

STUDY DESCRIPTION:

This is a single-arm prospective study to assess the feasibility, toxicity and cosmetic outcome of partial radiotherapy of the chest wall in breast cancer patients at increased risk of local relapse submitted to skin/nipple-areola complex (NAC) sparing mastectomy and immediate implant-based reconstruction

STUDY TYPE Interventional

STUDY DESIGN Endpoint Classification: Feasibility/Safety Study Intervention Model: Single Group Assignment Masking: Open Label Primary Purpose: Treatment

INCLUSION CRITERIA AND EXCLUSION CRITERIA (see below)

RADIOLOGY All patients will be submitted to preoperative full radiological work up including mammography, ultrasound scan and breast MRI in order to define precise tumor localization and extension (e.g. area covered by multiple tumor foci and/or extension of in situ associated to invasive tumor).

Immediately before surgery, non-permanent marks will be placed to delineate the skin covering the breast area involved by the tumor and two projection photographs will be taken and stored.

SURGERY NAC sparing or skin-sparing (in case of preoperative/intraoperative diagnosis of tumor involvement of the nipple ducts) mastectomy will be performed by raising thin skin flaps at the level of the superficial and deep fascia. The specimen will be oriented in the three dimensions by placement of stitches and sent for definitive pathology . The area of the pectoralis major muscle localized under the tumor will be delineated by placing 4 titanium radiopaque clips at cardinal points.

Nodal staging will be performed either by sentinel node biopsy, intraoperative evaluation and immediate/delayed full axillary dissection in case of macrometastatic sentinel node, or immediate full axillary dissection in case of preoperative citological diagnosis of metastatic axillary node.

RADIOTHERAPY The tumor bed is defined by the area at risk (skin and the pectoralis muscles) delineated by indelible skin marks (placed under the guidance of preoperative non-permanent skin marks) and surgical clips and 3D-MRI reconstruction for a precise localization of the tumor excised. The clinical target volume (CTV) is defined as the tumor bed with a 1.5 cm margin limited by skin contour.

The planning tumor volume (PTV) is defined using 4D-CT imaging and includes CTV plus 0.3/0.5 mm for setup error contribution. Internal target volume (ITV) accounts for motion of CTV in the patient.

Contouring of the target and organs at risk (OARs) is performed using both 3D-CT and 4D-CT imaging. All patients are scanned on a Aquilion Big Bore CT scanner (Toshiba). For generating 4D-CT datasets, a respiratory sensor box, integrated with the CT scanner reconstruction, is placed on the patient's chest. After the scan, the source data and the respiratory signal are used to retrospectively reconstruct the images. A maximum intensity projection (MIP) reconstruction over all respiratory phase is used to delineate target volumes. The contouring of OARs is performed using 3D-CT images.

Treatment plan is performed using Eclipse Treatment Planning System (TPS) or Tomotherapy TPS. Patients are treated with Volumetric Modulated Arc Therapy (VMAT) technique (1/2 half arcs) or helical Tomotherapy using 6 MV photon beams. Treatment plans is optimized for coverage and homogeneity. Clinically significant maximum target dose up to 112% is considered acceptable. A comparison plan using standard tangential fields is performed for each patient.

A dose of 40 Gy is delivered in 16 fractions (2.5 Gy per fraction). For conventional post-mastectomy radiotherapy this moderately hypofractionated schedule is considered feasible and safe (31). Even more so, this schedule should be feasible and safe for a smaller irradiated volume as in the current protocol. Regional nodal irradiation is not considered at our Institution for patients fulfilling the entry criteria of the protocol.

For patient setup verification, a cone-beam kVCT or a MVCT scan are performed before each treatment fraction and compared to the planning CT. Automatic registration between the reference and verification images is realised; patient position is corrected using a 6-degrees of freedom robotic couch top (linac) or a 4-degrees of freedom robotic couch top (Tomotherapy). Patients are immobilized using an arm shuttle device.

OUTCOME MEASURES PRIMARY

1. To assess the feasibility of PCWRT via VMAT-IGRT linac-based or helical Tomotherapy

   Surgical clips and permanent skin marks must allow proper identification of tumor bed both at CT imaging and on board imaging (CBCT-MVCT). The dose distribution must respect the standard dose constraints utilized in conventional CWRT. The following parameters will be evaluated:

   1.1. Patient set-up reproducibility 1.2. Plan reproducibility through in vivo dosimetry 1.3. Dosimetrical reduction of PCWRT vs. conventional CWRT
2. To assess the safety of PCWRT via VMAT-IGRT linac-based or helical Tomotherapy

   With hypofractionated CWRT the most frequent toxicity is acute skin toxicity (G2 skin toxicity in 10% of the cases). All toxicities are expected to be lower with PCWRT as compared to conventional CWRT since the radiation field is smaller. The following parameters will be evaluated:

   2.1. Acute and late cutaneous toxicity 2.2. Late subcutaneous fibrosis 2.3. Radiation pneumonitis
3. To assess the surgical complications of implant-based breast reconstruction after PCWRT

Reconstruction failures (RF), defined as the removal of the tissue expander/prosthesis, of conventional CWRT are reported in 20% of the cases. As for toxicities, also surgical complication rates are expected to be lower with PCWRT as compared to conventional CWRT since the radiation field of is smaller. The following parameters will be evaluated:

3.1. Infections, Skin/NAC necrosis, major revisions, early capsular contracture 3.2. Complication rates leading to implant removal.

SECONDARY

1. To assess the cosmetic outcome of implant-based breast reconstruction after PCWRT 1.1 An acceptable cosmetic result (excellent or good, on a scale of excellent-good-fair-poor) is defined as a stable reconstruction with good symmetry and contour relative to the contralateral breast.

   1.2 Outcome will be measured by means of photographic analysis using five views (frontal, right and left lateral, and right and left quarter views) and independent assessment of the results by a plastic surgeon who has not treated the patient.

   1.3 The modified Baker classification will be used to score the extent of contracture seen in the photographs
2. To assess patients' satisfaction of implant-based breast reconstruction after PCWRT 2.1 The BREAST-Q Reconstruction Module Patient Satisfaction with Breasts survey will be administered before and after treatment at predetermined time intervals

SAMPLE SIZE AND STATISTICAL CONSIDERATIONS No sample size calculation is appropriate because the main purpose of the proposed study is to assess the feasibility of PCWRT in order explore this intervention further in a large clinical trial.

Based on the clinical activity of the past 3 years at the Institute, 20 potential candidates per year are expected. If a 70% enrolment rate is hypothesized, a target accrual of 28 patients could be completed in two years. This target should allow to assess primary endpoint 1. appropriately and provide estimates of endpoints 2. and 3. that be used to design a subsequent larger clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of in situ ductal carcinoma (pTis) or invasive breast carcinoma (pT1 and pT2), submitted to NAC sparing mastectomy with prosthetic-based breast reconstruction (expander or prosthesis) and:
* Group A)

Negative sentinel node dissection or axillary clearance (pN0) and all the following risk factors:

* Close (less than 1 mm) or positive (ink on tumor margin) surgical margin in a single breast quadrant
* Tumor diameter >2 cm
* Age ≤50 years
* Grade 3 histology

  * Group B)

Positive sentinel dissection (pN1a) followed by axillary clearance (or primary axillary clearance) with only 1 positive node and any of the following risk factors:

* Close (less than 1 mm) or positive (ink on tumor margin) surgical margins in a single breast quadrant
* Age ≤50 years
* Tumor diameter >2 cm
* Grade 3 histology
* Lymphovascular invasion
* HER-2 overexpression/amplification
* Triple negativity

  * Patients must be older than 18 and less than 81 years of age
  * WHO (ECOG) Performance Status of 0-2
  * Patients must consent to return for scheduled treatments and follow up
  * Written informed consent document signed

Exclusion Criteria:

* Stages IIIB, IIIC and IV (any T4, any N3 or M1)
* Pathological metastasis in ≥2 axillary lymph nodes, clinically apparent metastasis in internal mammary and/or supraclavicular lymph nodes
* Close (less than 1 mm) or positive (ink on tumor margin) surgical margin in multiple breast quadrants
* Patients submitted to neoadjuvant chemotherapy
* Recurrence of breast cancer following mastectomy and/or adjuvant chemotherapy.
* Concomitant primary cancer in the contralateral breast
* History of other malignancy except carcinoma in situ of the cervix or non-melanoma skin cancer
* Pregnant or breast-feeding
* Other severe concomitant disease that could impact upon the ability to deliver treatment or increase the risk of toxicity (such as uncompensated congestive heart failure, unstable coronary heart disease, uncompensated chronic obstructive pulmonary disease, collagen vascular diseases including systemic lupus erythematosus, systemic sclerosis, dermatomyositis, and ataxia telangiectasia)
* Contraindications to radiation therapy (such as previous irradiation of the breast or chest wall)
* Severe psychiatric disorder that may interfere with the process of informed consent and/or treatment or follow-up compliance

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Assess feasibility , defined as patient set-up reproducibility, plan reproducibility through in vivo dosimetry and dosimetrical reduction of PCWRT vs. conventional chest wall radiotherapy | 5 weeks
  Evaluation of reproducibility of the technique. Evaluation of dose administered to non-target organ.

SECONDARY OUTCOMES:
Assess safety basing on RTOG ACUTE Radiation Morbidity and RTOG/EORTC LATE Radiation Morbidity | 6-24 months following the completion of radiation therapy
  Number of patients who developed toxicities on the treated chest wall, on the contralateral breast, on the lung, on the hearth. It will be evaluated also the grade of toxicities.
Assess surgical complication using a four-step scale of capsular contracture after prosthetic breast reconstruction | 6, 12, 18 and 24 months following the completion of radiation therapy
  Evaluation of early and late surgical complication as infection, skin necrosis, major revisions and capsular contraction
Assess cosmetic outcome using a qualitative scale (excellent-good-fair-poor) | 1, 3, 6, 12, 18 and 24 months following the completion of radiation therapy
  Evaluation of the quality of reconstruction defined as a stable reconstruction with good symmetry and contour relative to the contralateral breast
Assess patients' satisfaction throuhg a questionnaire administered to patients | 12 months following the completion of radiation therapy
  Evaluation of the perception of the patients about the outcome of prosthetic breast reconstruction

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Ponzone, MD, Principal Investigator — Fondazione del Piemonte per l'Oncologia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Recht A, Edge SB, Solin LJ, Robinson DS, Estabrook A, Fine RE, Fleming GF, Formenti S, Hudis C, Kirshner JJ, Krause DA, Kuske RR, Langer AS, Sledge GW Jr, Whelan TJ, Pfister DG; American Society of Clinical Oncology. Postmastectomy radiotherapy: clinical practice guidelines of the American Society of Clinical Oncology. J Clin Oncol. 2001 Mar 1;19(5):1539-69. doi: 10.1200/JCO.2001.19.5.1539. PMID 11230499
- [Background] EBCTCG (Early Breast Cancer Trialists' Collaborative Group); McGale P, Taylor C, Correa C, Cutter D, Duane F, Ewertz M, Gray R, Mannu G, Peto R, Whelan T, Wang Y, Wang Z, Darby S. Effect of radiotherapy after mastectomy and axillary surgery on 10-year recurrence and 20-year breast cancer mortality: meta-analysis of individual patient data for 8135 women in 22 randomised trials. Lancet. 2014 Jun 21;383(9935):2127-35. doi: 10.1016/S0140-6736(14)60488-8. Epub 2014 Mar 19. PMID 24656685
- [Background] Nordenskjold AE, Fohlin H, Albertsson P, Arnesson LG, Chamalidou C, Einbeigi Z, Holmberg E, Nordenskjold B, Karlsson P. No clear effect of postoperative radiotherapy on survival of breast cancer patients with one to three positive nodes: a population-based study. Ann Oncol. 2015 Jun;26(6):1149-1154. doi: 10.1093/annonc/mdv159. Epub 2015 Apr 3. PMID 25839671
- [Background] Karlsson P, Cole BF, Chua BH, Price KN, Lindtner J, Collins JP, Kovacs A, Thurlimann B, Crivellari D, Castiglione-Gertsch M, Forbes JF, Gelber RD, Goldhirsch A, Gruber G; International Breast Cancer Study Group. Patterns and risk factors for locoregional failures after mastectomy for breast cancer: an International Breast Cancer Study Group report. Ann Oncol. 2012 Nov;23(11):2852-2858. doi: 10.1093/annonc/mds118. Epub 2012 Jul 9. PMID 22776708
- [Background] Huo D, Hou N, Jaskowiak N, Winchester DJ, Winchester DP, Yao K. Use of Postmastectomy Radiotherapy and Survival Rates for Breast Cancer Patients with T1-T2 and One to Three Positive Lymph Nodes. Ann Surg Oncol. 2015 Dec;22(13):4295-304. doi: 10.1245/s10434-015-4528-x. Epub 2015 Mar 28. PMID 25820998
- [Background] Recht A, Comen EA, Fine RE, Fleming GF, Hardenbergh PH, Ho AY, Hudis CA, Hwang ES, Kirshner JJ, Morrow M, Salerno KE, Sledge GW Jr, Solin LJ, Spears PA, Whelan TJ, Somerfield MR, Edge SB. Postmastectomy Radiotherapy: An American Society of Clinical Oncology, American Society for Radiation Oncology, and Society of Surgical Oncology Focused Guideline Update. J Clin Oncol. 2016 Dec 20;34(36):4431-4442. doi: 10.1200/JCO.2016.69.1188. Epub 2016 Sep 30. PMID 27646947
- [Background] Budach W, Kammers K, Boelke E, Matuschek C. Adjuvant radiotherapy of regional lymph nodes in breast cancer - a meta-analysis of randomized trials. Radiat Oncol. 2013 Nov 14;8:267. doi: 10.1186/1748-717X-8-267. PMID 24225206
- [Background] Jagsi R, Raad RA, Goldberg S, Sullivan T, Michaelson J, Powell SN, Taghian AG. Locoregional recurrence rates and prognostic factors for failure in node-negative patients treated with mastectomy: implications for postmastectomy radiation. Int J Radiat Oncol Biol Phys. 2005 Jul 15;62(4):1035-9. doi: 10.1016/j.ijrobp.2004.12.014. PMID 15990006
- [Background] Abi-Raad R, Boutrus R, Wang R, Niemierko A, Macdonald S, Smith B, Taghian AG. Patterns and risk factors of locoregional recurrence in T1-T2 node negative breast cancer patients treated with mastectomy: implications for postmastectomy radiotherapy. Int J Radiat Oncol Biol Phys. 2011 Nov 1;81(3):e151-7. doi: 10.1016/j.ijrobp.2011.01.015. Epub 2011 Mar 21. PMID 21420245
- [Background] Ahlborn TN, Gump FE, Bodian C, Habif DV, Kister S. Tumor to fascia margin as a factor in local recurrence after modified radical mastectomy. Surg Gynecol Obstet. 1988 Jun;166(6):523-6. PMID 3375963
- [Background] Mentzer SJ, Osteen RT, Wilson RE. Local recurrence and the deep resection margin in carcinoma of the breast. Surg Gynecol Obstet. 1986 Dec;163(6):513-7. PMID 3024341
- [Background] Freedman GM, Fowble BL, Hanlon AL, Myint MA, Hoffman JP, Sigurdson ER, Eisenberg BL, Goldstein LJ, Fein DA. A close or positive margin after mastectomy is not an indication for chest wall irradiation except in women aged fifty or younger. Int J Radiat Oncol Biol Phys. 1998 Jun 1;41(3):599-605. doi: 10.1016/s0360-3016(98)00103-5. PMID 9635708
- [Background] Kunkler IH, Canney P, van Tienhoven G, Russell NS; MRC/EORTC (BIG 2-04) SUPREMO Trial Management Group. Elucidating the role of chest wall irradiation in 'intermediate-risk' breast cancer: the MRC/EORTC SUPREMO trial. Clin Oncol (R Coll Radiol). 2008 Feb;20(1):31-4. doi: 10.1016/j.clon.2007.10.004. No abstract available. PMID 18345543
- [Background] Jagsi R, Jiang J, Momoh AO, Alderman A, Giordano SH, Buchholz TA, Kronowitz SJ, Smith BD. Trends and variation in use of breast reconstruction in patients with breast cancer undergoing mastectomy in the United States. J Clin Oncol. 2014 Mar 20;32(9):919-26. doi: 10.1200/JCO.2013.52.2284. Epub 2014 Feb 18. PMID 24550418
- [Background] Mahmood U, Hanlon AL, Koshy M, Buras R, Chumsri S, Tkaczuk KH, Cheston SB, Regine WF, Feigenberg SJ. Increasing national mastectomy rates for the treatment of early stage breast cancer. Ann Surg Oncol. 2013 May;20(5):1436-43. doi: 10.1245/s10434-012-2732-5. Epub 2012 Nov 8. PMID 23135312
- [Background] Kummerow KL, Du L, Penson DF, Shyr Y, Hooks MA. Nationwide trends in mastectomy for early-stage breast cancer. JAMA Surg. 2015 Jan;150(1):9-16. doi: 10.1001/jamasurg.2014.2895. PMID 25408966
- [Background] Barry M, Kell MR. Radiotherapy and breast reconstruction: a meta-analysis. Breast Cancer Res Treat. 2011 May;127(1):15-22. doi: 10.1007/s10549-011-1401-x. Epub 2011 Feb 20. PMID 21336948
- [Background] Piper M, Peled AW, Foster RD, Moore DH, Esserman LJ. Total skin-sparing mastectomy: a systematic review of oncologic outcomes and postoperative complications. Ann Plast Surg. 2013 Apr;70(4):435-7. doi: 10.1097/SAP.0b013e31827e5333. PMID 23486127
- [Background] Weidong Li, Shuling Wang, Xiaojing Guo, Ronggang Lang, Yu Fan, Feng Gu, Xinmin Zhang, Zhengmao Zhu, Yun Niu, Li Fu. Nipple involvement in breast cancer: retrospective analysis of 2323 consecutive mastectomy specimens. Int J Surg Pathol. 2011 Jun;19(3):328-34. doi: 10.1177/1066896911399279. Epub 2011 Mar 31. PMID 21454374
- [Background] Rusby JE, Smith BL, Gui GP. Nipple-sparing mastectomy. Br J Surg. 2010 Mar;97(3):305-16. doi: 10.1002/bjs.6970. PMID 20101646
- [Background] De La Cruz L, Moody AM, Tappy EE, Blankenship SA, Hecht EM. Overall Survival, Disease-Free Survival, Local Recurrence, and Nipple-Areolar Recurrence in the Setting of Nipple-Sparing Mastectomy: A Meta-Analysis and Systematic Review. Ann Surg Oncol. 2015 Oct;22(10):3241-9. doi: 10.1245/s10434-015-4739-1. Epub 2015 Aug 5. PMID 26242363
- [Background] Agarwal S, Agarwal J. Radiation delivery in patients undergoing therapeutic nipple-sparing mastectomy. Ann Surg Oncol. 2015 Jan;22(1):46-51. doi: 10.1245/s10434-014-3932-y. Epub 2014 Jul 19. PMID 25037972
- [Background] Petit JY, Veronesi U, Orecchia R, Rey P, Martella S, Didier F, Viale G, Veronesi P, Luini A, Galimberti V, Bedolis R, Rietjens M, Garusi C, De Lorenzi F, Bosco R, Manconi A, Ivaldi GB, Youssef O. Nipple sparing mastectomy with nipple areola intraoperative radiotherapy: one thousand and one cases of a five years experience at the European institute of oncology of Milan (EIO). Breast Cancer Res Treat. 2009 Sep;117(2):333-8. doi: 10.1007/s10549-008-0304-y. Epub 2009 Jan 17. PMID 19152026
- [Background] Benediktsson KP, Perbeck L. Survival in breast cancer after nipple-sparing subcutaneous mastectomy and immediate reconstruction with implants: a prospective trial with 13 years median follow-up in 216 patients. Eur J Surg Oncol. 2008 Feb;34(2):143-8. doi: 10.1016/j.ejso.2007.06.010. Epub 2007 Aug 20. PMID 17709228
- [Background] Sakurai T, Zhang N, Suzuma T, Umemura T, Yoshimura G, Sakurai T, Yang Q. Long-term follow-up of nipple-sparing mastectomy without radiotherapy: a single center study at a Japanese institution. Med Oncol. 2013 Mar;30(1):481. doi: 10.1007/s12032-013-0481-3. Epub 2013 Feb 2. PMID 23377926
- [Background] Wilkinson JB, Beitsch PD, Shah C, Arthur D, Haffty BG, Wazer DE, Keisch M, Shaitelman SF, Lyden M, Chen PY, Vicini FA. Evaluation of current consensus statement recommendations for accelerated partial breast irradiation: a pooled analysis of William Beaumont Hospital and American Society of Breast Surgeon MammoSite Registry Trial Data. Int J Radiat Oncol Biol Phys. 2013 Apr 1;85(5):1179-85. doi: 10.1016/j.ijrobp.2012.10.010. Epub 2012 Nov 22. PMID 23182700
- [Background] Klein J, Kong I, Paszat L, Nofech-Mozes S, Hanna W, Thiruchelvam D, Narod SA, Saskin R, Done SJ, Miller N, Youngson B, Tuck A, Sengupta S, Elavathil L, Jani PA, Slodkowska E, Bonin M, Rakovitch E. Close or positive resection margins are not associated with an increased risk of chest wall recurrence in women with DCIS treated by mastectomy: a population-based analysis. Springerplus. 2015 Jul 10;4:335. doi: 10.1186/s40064-015-1032-5. eCollection 2015. PMID 26185737
- [Background] Ponzone R, Maggiorotto F, Carabalona S, Rivolin A, Pisacane A, Kubatzki F, Renditore S, Carlucci S, Sgandurra P, Marocco F, Magistris A, Regge D, Martincich L. MRI and intraoperative pathology to predict nipple-areola complex (NAC) involvement in patients undergoing NAC-sparing mastectomy. Eur J Cancer. 2015 Sep;51(14):1882-9. doi: 10.1016/j.ejca.2015.07.001. Epub 2015 Jul 22. PMID 26210374
- [Background] Vaidya JS, Wenz F, Bulsara M, Tobias JS, Joseph DJ, Keshtgar M, Flyger HL, Massarut S, Alvarado M, Saunders C, Eiermann W, Metaxas M, Sperk E, Sutterlin M, Brown D, Esserman L, Roncadin M, Thompson A, Dewar JA, Holtveg HM, Pigorsch S, Falzon M, Harris E, Matthews A, Brew-Graves C, Potyka I, Corica T, Williams NR, Baum M; TARGIT trialists' group. Risk-adapted targeted intraoperative radiotherapy versus whole-breast radiotherapy for breast cancer: 5-year results for local control and overall survival from the TARGIT-A randomised trial. Lancet. 2014 Feb 15;383(9917):603-13. doi: 10.1016/S0140-6736(13)61950-9. Epub 2013 Nov 11. PMID 24224997
- [Background] Gatti M, Ponzone R, Bresciani S, Panaia R, Kubatzki F, Maggiorotto F, Di Virgilio MR, Salatino A, Baiotto B, Montemurro F, Stasi M, Gabriele P. Accelerated partial breast irradiation using 3D conformal radiotherapy: toxicity and cosmetic outcome. Breast. 2013 Dec;22(6):1136-41. doi: 10.1016/j.breast.2013.07.042. Epub 2013 Aug 16. PMID 23958374
- [Background] Ko DH, Norriss A, Harrington CR, Robinson BA, James ML. Hypofractionated radiation treatment following mastectomy in early breast cancer: the Christchurch experience. J Med Imaging Radiat Oncol. 2015 Apr;59(2):243-7. doi: 10.1111/1754-9485.12242. Epub 2014 Oct 6. PMID 25287654
- [Background] Billingham SA, Whitehead AL, Julious SA. An audit of sample sizes for pilot and feasibility trials being undertaken in the United Kingdom registered in the United Kingdom Clinical Research Network database. BMC Med Res Methodol. 2013 Aug 20;13:104. doi: 10.1186/1471-2288-13-104. PMID 23961782
- [Background] Momoh AO, Ahmed R, Kelley BP, Aliu O, Kidwell KM, Kozlow JH, Chung KC. A systematic review of complications of implant-based breast reconstruction with prereconstruction and postreconstruction radiotherapy. Ann Surg Oncol. 2014 Jan;21(1):118-24. doi: 10.1245/s10434-013-3284-z. Epub 2013 Oct 1. PMID 24081801